CLINICAL TRIAL: NCT02116543
Title: A Double-Blinded, Randomized, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Antiviral Activity of TD-6450, a NS5A Inhibitor, in Treatment Naïve Subjects With Genotype 1, 2 or 3 Chronic Hepatitis C Virus (HCV)
Brief Title: TD-6450 MAD Study in HCV Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0110
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C; HCV
Keywords: Hepatitis C; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-6450 (Experimental): TD-6450 capsules
  Interventions: Drug: TD-6450
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-6450
  Arms: TD-6450
Drug: Placebo
  Arms: Placebo

SUMMARY:
This proof of concept study is designed to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of TD-6450 in treatment naïve subjects with GT-1, GT-2 or GT-3 chronic HCV.

ELIGIBILITY:
Inclusion Criteria:

* Subject is HCV antibody positive
* Subject is treatment naïve, with no history of exposure (single or multiple dose) to interferon, ribavirin or direct acting antivirals.
* Subject has had a liver biopsy within 3 years or Fibroscan evaluation within 6 months prior to Screening that clearly excludes cirrhosis. If not available prior to Screening, the absence of cirrhosis must be confirmed prior to subject enrollment using either Fibroscan or Fibrosure®.
* Subject is negative for hepatitis A (HAV), hepatitis B (HBV), and human immunodeficiency virus (HIV).

Exclusion Criteria:

* Subject has prior histological evidence of cirrhosis or current clinical evidence of cirrhosis in the opinion of the investigator.
* Subject has a history or evidence of non-hepatitis C chronic liver disease.
* Subject has an estimated creatinine clearance of <80 ml/min if 18-60 years of age, inclusive; or <70 ml/min if >60 years of age, calculated using the Cockcroft-Gault equation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | 28 Days
  Number, type, severity, and association of treatment emergent adverse events.

SECONDARY OUTCOMES:
Cmax | 28 Days
  Cmax
Tmax | 28 Days
  Tmax
AUC0-t | 28 Days
AUC0-∞ | 28 Days
  AUC0-∞
AUC0-24 | 28 Days
Antiviral Activity | 28 Days
  Change from baseline in HCV RNA
t1/2 | 28 Days
  t1/2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Texas Liver Institute, San Antonio, Texas, United States